CLINICAL TRIAL: NCT01436799
Title: International Review Board of Gachon University Gil Hospital
Brief Title: Desflurane Versus Propofol in the Sitting Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Hyun Jeong Kwak, Associate professor, Gachon University Gil Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GIRBA2466
Record Dates: First submitted 2011-09-15; First posted 2011-09-20 (Estimated); Results first posted 2013-08-26 (Estimated); Last update posted 2013-09-09 (Estimated); Status verified 2013-08

CONDITIONS: Cerebral Ischemia
Keywords: propofol; desflurane; cerebrovascular circulation; sitting
MeSH Terms: conditions — Brain Ischemia | interventions — Propofol; Desflurane; Desmin; Alfentanil; GTF2A1L protein, human; Rocuronium; ROC Curve

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Desflurane (Experimental): anaesthesia was induced with thiopental sodium 2 mg kg-1, alfentanil 10 μg kg-1 and rocuronium 0.6 mg kg-1. Anesthetic maintenance by desflurane
  Interventions: Drug: Desflurane; Drug: alfentanil; Drug: Rocuronium
- propofol (Active Comparator): anaesthesia was induced with the effect-site concentration of propofol 5.0 μg ml-1, alfentanil 10 μg kg-1, and rocuronium 0.6 mg kg-1. A commercially available target controlled infusion (TCI) pump (Orchestra®, Fresenius Vial, France) was used and the pharmacokinetic set used to calculate target effect-site concentrations for propofol was Schnider and colleagues' model
  Interventions: Drug: propofol; Drug: alfentanil; Drug: Rocuronium

INTERVENTIONS:
Drug: propofol — anaesthesia was induced with the effect-site concentration of propofol 5.0 μg ml-1 mainly.
  Arms: propofol
Drug: Desflurane — anaesthesia was maintained by desflurane 4-7vol%
  Other Names: Des
  Arms: Desflurane
Drug: alfentanil — administration of alfentanil 10 μg kg-1 for anesthetic induction
  Other Names: alf
Drug: Rocuronium — administration of rocuronium 0.6 mg kg-1 for anesthetic induction
  Other Names: roc

SUMMARY:
The investigators hypothesized that both propofol and desflurane would decrease the regional oxygen saturation (rSO2) but propofol is likely to reduce rSO2 more than sevoflurane when patients are raised to the sitting position.

DETAILED DESCRIPTION:
The investigators hypothesized that both propofol and desflurane would decrease the rSO2 but propofol is likely to reduce rSO2 more than sevoflurane when patients are raised to the sitting position. Therefore, the purpose of this study was to investigate the effect of desflurane and propofol on rSO2 values during the beach chair position for shoulder arthroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Forty patients,
* ASA class I or II,
* undergoing shoulder arthroscopy

Exclusion Criteria:

* Patients with history of cerebrovascular disease, coronary occlusive disease and/or obesity (body mass index > 30) were excluded from this study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-03; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Jeong Kwak, MD.PhD, Study Director — Gachon University Gil Medical Center

RESULTS

PARTICIPANT FLOW:
Recruitment Details: March 2011-August 2011 in Gachon University Gil Medical Center, who underwent arthroscopic shoulder surgery
Pre-assignment Details: no enrolled participants were excluded.
Period: Overall Study
Arm/Group | Desflurane | Propofol
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Desflurane | Propofol | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 48 (10) | 48 (16) | 48 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 11 | 14 | 25
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Regional Cerebral Oxygen Satuation (rSO2)
Description: definitive values of regional cerebral oxygen saturation(rSO2,%) values are described as mean (SD)
Time Frame: 1, 3, 5, 7, and 9 min after the beach chair position
Population: A power analysis was calculated based on a previous study.14 In each group, 16 patients were needed to detect a mean intergroup difference of 5% in the rSO2 value with a power of 80% and a type I error of 0.05. To compensate for a dropout rate of 20%, 40 patients were included in this study.
Measure: Mean (Standard Deviation); unit: percentage of rSO2 (%)
Groups:
- Desflurane: anesthetic maintenence with desflurane
- Propofol: anesthetic maintanence with propofol
Arm/Group | Desflurane | Propofol
Number analyzed (Participants) | 20 | 20
percentage of rSO2 (%)
  1min after beach chair position | 77.4 (7) | 72.5 (9.5)
  3min after beach chair position | 76 (7.1) | 70 (9.8)
  5min after beach chair position | 75.2 (7.4) | 70 (8.5)
  7min after beach chair position | 75.1 (7.2) | 68.5 (10.1)
  9min after beach chair position | 74 (7.8) | 67.8 (9.8)

ADVERSE EVENTS:
Time Frame: 1, 3, 5, 7 and 9 min after the sitting position and postoperative 24hours
Arm/Group | Desflurane | Propofol
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
limitations of this study is that the ventilation was adjusted according to ETCO2 value instead of the arterial carbon dioxide tensions (PaCO2).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No